CLINICAL TRIAL: NCT03456700
Title: Phase II Trial to Evaluate the Efficacy of Auranofin and Sirolimus in Serous Ovarian Cancer Patients With Recurrent Disease
Brief Title: Auranofin and Sirolimus in Treating Participants With Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is closed per results from the interim analysis.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1761; NCI-2018-00321 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1761 (Other: Mayo Clinic); 17-005302 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Serous Tumor; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Auranofin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (auranofin, sirolimus) (Experimental): Participants receive auranofin PO QD and sirolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Auranofin; Other: Laboratory Biomarker Analysis; Drug: Sirolimus

INTERVENTIONS:
Drug: Auranofin — Given PO
  Other Names: Ridaura
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217

SUMMARY:
This phase II trial studies how well auranofin and sirolimus work in treating participants with ovarian cancer. Immunosuppressive therapy, such as auranofin and sirolimus, is used to decrease the body?s immune response and may increase blood cell count.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall tumor response rate (ORR, that is, complete response [CR] + partial response [PR]) of the combination of auranofin and sirolimus in the setting of metastatic serous ovarian cancer across all patients.

SECONDARY OBJECTIVES:

I. To estimate the overall tumor response rate (ORR, that is, complete response [CR] + partial response [PR]) of the combination of auranofin and sirolimus in the setting of metastatic serous ovarian cancer within patients that have overexpression of PKCiota.

II. To estimate progression-free survival, overall survival, and adverse events from the combination of auranofin and sirolimus.

CORRELATIVE OBJECTIVES:

I. To explore whether PKCiota-relevant biomarkers in serous ovarian cancer tumors are associated with treatment response patterns, such as ORR, progression free survival, and overall survival.

OUTLINE:

Participants receive auranofin orally (PO) once daily (QD) and sirolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, participants are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Ovarian, Fallopian Tube or Primary Peritoneal cancer of serous histology
* Incurable cancer
* Willingness to provide paraffin-embedded tissue blocks of ovarian cancer
* Measurable disease
* Obtained =< 14 days prior to registration: Absolute neutrophil count (ANC) >= 1500 uL
* Obtained =< 14 days prior to registration: Platelet (PLT) >= 100,000 uL
* Obtained =< 14 days prior to registration: Hemoglobin (Hgb) >= 9 g/dL
* Obtained =< 14 days prior to registration: Total bilirubin =< 1.5 x upper limit of normal (ULN) or direct bilirubin =< ULN
* Obtained =< 14 days prior to registration: Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN or SGOT (AST) and SGPT (ALT) =< 5 x ULN is acceptable if liver has tumor involvement
* Obtained =< 14 days prior to registration: Creatinine =< 1.5 x ULN
* Obtained =< 14 days prior to registration: Fasting serum glucose =< 1.5 x ULN
* Obtained =< 14 days prior to registration: Total cholesterol =< 1.5 x ULN
* Obtained =< 14 days prior to registration: Triglycerides =< 1.5 x ULN
* Life expectancy >= 12 weeks

Exclusion Criteria:

* Platinum-sensitive disease (exceptions allowed: patient has had a hypersensitivity reaction to platinum or the treating oncologist thinks that further platinum therapy is not in the patient?s best interest)
* Morbidities or concurrent major illness (for example, bowel obstruction or a second active malignancy) that, in the opinion of the treating healthcare provider, would make participation in the trial problematic
* Leptomeningeal disease or uncontrolled brain metastasis
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment

  * NOTE: Patients can have peripheral (sensory) neuropathy
* History of hypertriglyceridemia or hypercholesterolemia and currently on medication(s)
* Use of St. John?s wort =< 7 days prior to registration
* Unable to discontinue use of a strong CYP3A4 inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Jatoi A, Foster NR, Wahner Hendrickson A, Block MS, Weroha SJ, Asmus EJ, Murray NR, Fields AP. A Phase 2 Trial of Protein Kinase C Iota Inhibition With the Combination of Auranofin and Sirolimus in Patients With Recurrent Ovarian Cancer. Am J Clin Oncol. 2025 Oct 20. doi: 10.1097/COC.0000000000001263. Online ahead of print. PMID 41114938
- [Derived] Rousselle B, Massot A, Privat M, Dondaine L, Trommenschlager A, Bouyer F, Bayardon J, Ghiringhelli F, Bettaieb A, Goze C, Paul C, Malacea-Kabbara R, Bodio E. Conception and Evaluation of Fluorescent Phosphine-Gold Complexes: From Synthesis to in vivo Investigations. ChemMedChem. 2022 Jun 3;17(11):e202100773. doi: 10.1002/cmdc.202100773. Epub 2022 Mar 29. PMID 35254001
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Auranofin, Sirolimus): Participants receive 6 mg auranofin PO QD and 5 mg sirolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
Period: Overall Study
Arm/Group | Treatment (Auranofin, Sirolimus)
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Received prior chemotherapy for this cancer [Count of Participants; unit: Participants] | 20
Tumor Over-expression of Protein Kinase C (PKC) iota [Count of Participants; unit: Participants] | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Confirmed Tumor Response (Partial Response [PR] or Complete Response [CR] at Least 4 Weeks Apart)
Description: The outcome measure is the number of participants with a confirmed tumor response (partial response [PR] or complete response [CR] at least 4 weeks apart). PR and CR are defined using RECIST 1.1 criteria. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR: Disappearance of all target and non-target lesions and normalisation of tumour marker level. Any pathological lymph nodes must have reduction in short axis to <10 mm.
Time Frame: 1 year 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Number of Participants With a Confirmed Tumor Response (PR or CR at Least 4 Weeks Apart) in the Subset of Participants That Have Over-expression of Protein Kinase C (PKC) Iota
Description: The outcome measure is the number of participants with a confirmed tumor response (partial response [PR] or complete response [CR] at least 4 weeks apart) in the subset of participants that have overexpression of PKC iota. PR and CR are defined using RECIST 1.1 criteria. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR: Disappearance of all target and non-target lesions and normalisation of tumour marker level. Any pathological lymph nodes must have reduction in short axis to <10 mm.
Time Frame: 1 year 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
Participants | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from registration to the first of either disease progression or death from any cause. Patients who receive the study drug, but then never return for an evaluation will be censored on their last follow-up date. PFS will be estimated using the method of Kaplan-Meier. Progression is defined using RECIST 1.1 criteria; Progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression), Unequivocal progression (see comments below) of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered progression), or appearance of new malignant lesions.
Time Frame: 1 year 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
months | 2.1 [1.8 to 3.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from registration to death from any cause. OS will be estimated using the method of Kaplan-Meier.
Time Frame: 1 year 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
months | 4.4 [2.6 to 12.5]

5. Secondary Outcome: Number of Participants Experiencing at Least One Grade 3 or Worse Adverse Event (AE)
Description: The outcome measure is the number of participants experiencing at least one grade 3 or worse adverse event (AE).
Time Frame: 1 year 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Auranofin, Sirolimus)
Number analyzed (Participants) | 21
Participants | 13

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Participants evaluable for adverse events are summarized below (i.e. participants who did not withdraw consent).
Arm/Group | Treatment (Auranofin, Sirolimus)
All-Cause Mortality (participants affected / at risk) | 19/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Auranofin, Sirolimus) (N=21)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Auranofin, Sirolimus) (N=21)
Anemia (Blood and lymphatic system disorders) | 16 (26)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 17 (32)
Mucositis oral (Gastrointestinal disorders) | 12 (20)
Nausea (Gastrointestinal disorders) | 11 (17)
Vomiting (Gastrointestinal disorders) | 9 (12)
Edema limbs (General disorders) | 3 (5)
Fatigue (General disorders) | 19 (40)
Alkaline phosphatase increased (Investigations) | 2 (3)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 7 (12)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 6 (12)
White blood cell decreased (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (12)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 8 (13)
Proteinuria (Renal and urinary disorders) | 11 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03456700/Prot_SAP_000.pdf